CLINICAL TRIAL: NCT02620579
Title: Biopsychosocial Influence on Shoulder Pain: a Randomized, Pre-clinical Trial
Brief Title: Biopsychosocial Influence on Shoulder Pain
Acronym: BISP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00078287; 2R01AR055899 (NIH)
Record Dates: First submitted 2015-11-13; First posted 2015-12-03 (Estimated); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Shoulder Pain
Keywords: Personalized Pharmaceutical; Personalized Education
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Personalized Pharmaceutical and Education (Experimental): This group will have propranolol (Propranolol LA) 60 mg administered orally and receive the pain processing education modules as the combined intervention for this arm.
  Interventions: Drug: Propranolol LA (60 mg); Behavioral: Pain Processing Education
- Placebo Pharmaceutical, General Education (Placebo Comparator): This group will have the placebo pharmaceutical administered orally and receive general shoulder anatomy education modules as the interventions for this arm.
  Interventions: Drug: Placebo; Behavioral: Shoulder Anatomy Education
- Placebo Pharmaceutical, Personalized Education (Active Comparator): This group will have the placebo pharmaceutical administered orally and receive the pain processing education modules as the combined intervention for this arm.
  Interventions: Drug: Placebo; Behavioral: Pain Processing Education
- Personalized Pharmaceutical, General Education (Active Comparator): This group will have propranolol (Propranolol LA) 60 mg administered orally and receive general shoulder anatomy education modules as the interventions for this arm.
  Interventions: Drug: Propranolol LA (60 mg); Behavioral: Shoulder Anatomy Education

INTERVENTIONS:
Drug: Propranolol LA (60 mg) — Long-acting propranolol (Propranolol LA) 60 mg to be administered orally daily for Days 1 (before exercise induced muscle injury) and Days 2-4 following exercise induced muscle injury.
  Other Names: Personalized Pharmaceutical
  Arms: Personalized Pharmaceutical and Education; Personalized Pharmaceutical, General Education
Drug: Placebo — Placebo capsules will be prepared by the University of Florida Investigational Drug Service to be visually indistinguishable from the active medication and delivered orally. Placebo administration will be done in the same fashion as propranolol - administered on Days 1 (before exercise induced muscle injury) and the Days 2-4 after the exercise induced muscle injury.
  Other Names: Placebo Pharmaceutical
  Arms: Placebo Pharmaceutical, General Education; Placebo Pharmaceutical, Personalized Education
Behavioral: Shoulder Anatomy Education — Shoulder anatomy education modules will be administered Days 2-4 (after exercised induced muscle injury) following exercise enhance injury with the goal of participant understanding shoulder anatomy and injury while reviewing: a) structure and arthrokinematics of the shoulder joint; b) muscle anatomy of the shoulder with emphasis on the rotator cuff; and c) potential shoulder pain generators from the exercise-induced injury. This education component will be devoid of information related to pain signaling and cognitive restructuring that characterizes Pain Processing Education modules. These education modules will be scripted and structured so they are provided in a standardized manner for all subjects.
  Other Names: General Education
  Arms: Personalized Pharmaceutical, General Education; Placebo Pharmaceutical, General Education
Behavioral: Pain Processing Education — Pain processing education modules will be administered Days 2-4 (after exercised induced muscle injury) following exercise enhance injury with the goal of better understanding of pain processing and psycho-education. This information will encourage shoulder activation by: a) reducing the threat of muscle injury; b) encouraging normal use of the shoulder and arm; and c) addressing specific concerns expressed by the subject (e.g. pain with shoulder motion is a sign of re-injury). This education component will be devoid of detailed information on shoulder anatomy, movement, and injury that characterizes the Shoulder Anatomy Education modules. These education modules will be scripted and structured so they are provided in a standardized manner for all subjects.
  Other Names: Personalized Education
  Arms: Personalized Pharmaceutical and Education; Placebo Pharmaceutical, Personalized Education

SUMMARY:
Chronic shoulder pain is a common, costly, and disabling problem for society. The identification of factors predictive of the development of chronic shoulder pain is necessary to develop innovative and effective treatments to reduce the societal impact of shoulder disorders. In previous work the investigators identified a genetic and psychological subgroup that robustly predicted heightened shoulder pain responses in a pre-clinical cohort and poor 12 month shoulder pain recovery rates in a clinical surgical cohort. In this follow-up study the investigator proposes to test how interventions tailored to the high risk subgroup affect pain responses in a pre-clinical cohort.

The optimal theorized match for the identified high-risk subgroup is a combination of personalized pharmaceutical and education interventions. This combined personalized intervention versus a placebo pharmaceutical and general education intervention group is the primary comparison of interest. Also, an evaluation of the individual effect of personalized pharmaceutical and educational interventions will be part of the study. Such comparisons will provide important information on what the active portion of the combined personalized intervention may be.

DETAILED DESCRIPTION:
Potential subjects will be screened and those meeting the high-risk criteria based on COMT genotype for high pain sensitivity and pain catastrophizing questionnaire score will be eligible for randomization into intervention groups (stratified by sex). Exercise induced shoulder injury will serve as the pain generating mechanism on Day 1 and participants will receive pharmaceutical and education interventions over Days 1-4, and Days 2-4 respectively. Statistical analysis will determine whether the combined personalized intervention group experienced shorter shoulder pain duration, lower peak pain intensity, or decreased upper-extremity disability and determine which molecular, psychological, and pain sensitivity regulation mechanisms are associated with pain relief. A preliminary analysis is planned after the first 300 subjects are equally randomized to the 4 intervention groups. The comparison of interest for the preliminary analysis is the combined personalized intervention group with the placebo and general education group for the primary outcome. Depending on the results of this preliminary analysis the randomization pattern may change, with details of these changes available in the protocol paper.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

* chronic pain (> 3 months) in any area,
* currently experiencing neck or shoulder pain,
* previous history of neck or shoulder pain (operationally defined as experiencing neck or shoulder pain for longer than 48 hours or seeking medical treatment for neck or shoulder pain),
* neurological impairment of the in the upper-extremity (determined by loss of sensation, muscle weakness, and reflex changes),
* regular participation in upper-extremity weight training,
* currently or regular use of pain medication, and
* previous history of upper-extremity surgery.

Additional exclusion criteria for propranolol administration are reported history of or presence of any of the following cardiovascular conditions:

* clinically significant abnormal 12-lead ECG,
* sinus bradycardia (resting heart rate below 55 beats per minute),
* greater than first degree heart block,
* cardiac failure,
* coronary artery disease,
* uncontrolled hypertension (resting systolic blood pressure above 140 mm Hg), or hypotension (resting systolic blood pressure below 90 mm Hg),
* Wolff-Parkinson-White syndrome.

Non-cardiovascular reasons for study exclusion include:

* bronchial asthma,
* nonallergic bronchospasm,
* history of recent major surgery requiring general anesthesia,
* diabetes,
* pregnancy,
* major depression.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bishop, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical and Translational Science Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George SZ, Staud R, Borsa PA, Wu SS, Wallace MR, Greenfield WH, Mackie LN, Fillingim RB. Biopsychosocial influence on shoulder pain: Rationale and protocol for a pre-clinical trial. Contemp Clin Trials. 2017 May;56:9-17. doi: 10.1016/j.cct.2017.03.005. Epub 2017 Mar 14. PMID 28315479
- [Background] Borsa PA, Parr JJ, Wallace MR, Wu SS, Dai Y, Fillingim RB, George SZ. Genetic and psychological factors interact to predict physical impairment phenotypes following exercise-induced shoulder injury. J Pain Res. 2018 Oct 23;11:2497-2508. doi: 10.2147/JPR.S171498. eCollection 2018. PMID 30425562
- [Background] Butera KA, George SZ, Borsa PA, Dover GC. Prolonged Reduction in Shoulder Strength after Transcutaneous Electrical Nerve Stimulation Treatment of Exercise-Induced Acute Muscle Pain. Pain Pract. 2018 Nov;18(8):954-968. doi: 10.1111/papr.12690. Epub 2018 Apr 6. PMID 29505689
- [Derived] George SZ, Bishop MD, Wu SS, Staud R, Borsa PA, Wallace MR, Greenfield WH 3rd, Dai Y, Fillingim RB. Biopsychosocial influence on shoulder pain: results from a randomized preclinical trial of exercise-induced muscle injury. Pain. 2023 Feb 1;164(2):305-315. doi: 10.1097/j.pain.0000000000002700. Epub 2022 May 23. PMID 35604152
- See also: Abstract for citation and access to paper — https://www.ncbi.nlm.nih.gov/pubmed/28315479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Periodic screenings of volunteers were completed on the University of Florida campus and in the local community. All participants provided informed consent to screening. Participants who screened as being in the high-risk subgroup and appropriate for exercise-induced muscle injury were eligible for participation in the clinical trial and provided additional informed consent.
Pre-assignment Details: Participants who were eligible based on being in the high-risk subgroup and appropriate for exercise-induced muscle injury were required to take additional testing to determine the appropriateness of receiving propranolol and also identifying other medical reasons for exclusion. 3 enrolled participants were excluded/withdrawn pre-randomization.
Groups:
- Personalized Pharmaceutical and Education (C): This group will have propranolol (Propranolol LA) 60 mg administered orally and receive the pain processing education modules as the combined intervention for this arm.
  Propranolol LA (60 mg): Long-acting propranolol (Propranolol LA) 60 mg to be administered orally daily for Days 1 (before exercise induced muscle injury) and Days 2-4 following exercise induced muscle injury.
  Pain Processing Education: Pain processing education modules will be administered Days 2-4 (after exercised induced muscle injury) following exercise enhance injury with the goal of better understanding of pain processing and psycho-education. This information will encourage shoulder activation by: a) reducing the threat of muscle injury; b) encouraging normal use of the shoulder and arm; and c) addressing specific concerns expressed by the subject (e.g. pain with shoulder motion is a sign of re-injury). This education component will be devoid of detailed information on shoulder anatomy, movement, and injury that characterizes the Shoulder Anatomy Education modules. These education modules will be scripted and structured so they are provided in a standardized manner for all subjects.
- Placebo Pharmaceutical, General Education (B): This group will have the placebo pharmaceutical administered orally and receive general shoulder anatomy education modules as the interventions for this arm.
  Placebo: Placebo capsules will be prepared by the University of Florida Investigational Drug Service to be visually indistinguishable from the active medication and delivered orally. Placebo administration will be done in the same fashion as propranolol - administered on Days 1 (before exercise induced muscle injury) and the Days 2-4 after the exercise induced muscle injury.
  Shoulder Anatomy Education: Shoulder anatomy education modules will be administered Days 2-4 (after exercised induced muscle injury) following exercise enhance injury with the goal of participant understanding shoulder anatomy and injury while reviewing: a) structure and arthrokinematics of the shoulder joint; b) muscle anatomy of the shoulder with emphasis on the rotator cuff; and c) potential shoulder pain generators from the exercise-induced injury. This education component will be devoid of information related to pain signaling and cognitive restructuring that characterizes Pain Processing Education modules. These education modules will be scripted and structured so they are provided in a standardized manner for all subjects.
- Placebo Pharmaceutical, Personalized Education (A): This group will have the placebo pharmaceutical administered orally and receive the pain processing education modules as the combined intervention for this arm.
  Placebo: Placebo capsules will be prepared by the University of Florida Investigational Drug Service to be visually indistinguishable from the active medication and delivered orally. Placebo administration will be done in the same fashion as propranolol - administered on Days 1 (before exercise induced muscle injury) and the Days 2-4 after the exercise induced muscle injury.
  Pain Processing Education: Pain processing education modules will be administered Days 2-4 (after exercised induced muscle injury) following exercise enhance injury with the goal of better understanding of pain processing and psycho-education. This information will encourage shoulder activation by: a) reducing the threat of muscle injury; b) encouraging normal use of the shoulder and arm; and c) addressing specific concerns expressed by the subject (e.g. pain with shoulder motion is a sign of re-injury). This education component will be devoid of detailed information on shoulder anatomy, movement, and injury that characterizes the Shoulder Anatomy Education modules. These education modules will be scripted and structured so they are provided in a standardized manner for all subjects.
- Personalized Pharmaceutical, General Education (D): This group will have propranolol (Propranolol LA) 60 mg administered orally and receive general shoulder anatomy education modules as the interventions for this arm.
  Propranolol LA (60 mg): Long-acting propranolol (Propranolol LA) 60 mg to be administered orally daily for Days 1 (before exercise induced muscle injury) and Days 2-4 following exercise induced muscle injury.
  Shoulder Anatomy Education: Shoulder anatomy education modules will be administered Days 2-4 (after exercised induced muscle injury) following exercise enhance injury with the goal of participant understanding shoulder anatomy and injury while reviewing: a) structure and arthrokinematics of the shoulder joint; b) muscle anatomy of the shoulder with emphasis on the rotator cuff; and c) potential shoulder pain generators from the exercise-induced injury. This education component will be devoid of information related to pain signaling and cognitive restructuring that characterizes Pain Processing Education modules. These education modules will be scripted and structured so they are provided in a standardized manner for all subjects.
Period: Overall Study
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D)
Started | 62 | 57 | 57 | 57
Completed | 62 | 56 | 56 | 56
Not Completed | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population consists of 233 participants. 28 out of 261 randomized participants were excluded due to criteria related to the safety of propranolol administration (eg, abnormal ECG findings) or a candidate not being able to complete the study (eg, change in time commitment). These post-randomization exclusions were made for safety reasons and participants were excluded prior to any baseline data collection, induction of exercise-induced muscle injury, and treatment allocation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D) | Total
Number analyzed (Participants) | 62 | 57 | 57 | 57 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (5.3) | 20.3 (2.5) | 21.7 (5.9) | 20.5 (1.9) | 21.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 39 | 37 | 153
  Male | 22 | 20 | 18 | 20 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 14 | 19 | 21 | 77
  Not Hispanic or Latino | 39 | 43 | 38 | 36 | 156
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 15 | 20 | 18 | 18 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 10 | 15 | 13 | 7 | 45
  White | 33 | 20 | 24 | 31 | 108
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 0 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 57 | 57 | 57 | 233
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (4.4) | 23.9 (4.1) | 24.1 (4.5) | 23.4 (4.3) | 23.7 (4.3)
Fear of Pain Questionnaire (FPQ) [Mean (Standard Deviation); unit: units on a scale] — The Fear of Pain Questionnaire (FPQ) is a self-report instrument that was developed specifically to assess fear of different stimuli usually causing pain. FPQ ranges from 0 to 31 and higher scores indicate higher levels of fear.
  units on a scale | 14.5 (6.0) | 14.6 (7.0) | 15.6 (6.8) | 14.5 (5.5) | 14.8 (6.3)
Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking. PCS ranges from 0 to 34 and higher scores are associated with higher amounts of pain catastrophizing.
  units on a scale | 12.6 (9.1) | 12.6 (7.2) | 12.7 (9.0) | 11.4 (7.8) | 12.3 (8.3)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 (Patient Health Questionnaire-9) objectifies and assesses degree of depression severity via questionnaire. PDQ-9 ranges from 0 to 24 and higher scores indicate greater depression.
  units on a scale | 1.9 (2.3) | 2.8 (3.1) | 3.2 (4.4) | 2.9 (3.8) | 2.7 (3.5)
Tampa Scale for Kinesiophobia-11 (TSK-11) [Mean (Standard Deviation); unit: units on a scale] — Tampa Scale of Kinesiophobia (TSK) is an instrument for assessing fear-avoidance, fear of work-related activities, fear of movement, and fear of re-injury. TSK-11 is a shortened version. TSK-11 ranges from 0 to 42 and higher scores indicate greater kinesiophobia.
  units on a scale | 19.6 (4.7) | 19.5 (5.0) | 19.4 (5.7) | 19.8 (5.2) | 19.5 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Met the Recovery Criterion for Shoulder Pain Intensity
Description: The outcome has a range between 0 and 1, the higher scores mean a better outcome. Successful recovery was determined based on meeting the recovery criterion for shoulder pain intensity by at least 6 days. Specifically, recovery (Yes or No) was defined using Brief Pain Inventory (BPI) ratings as a current pain intensity rating of 0/10 and a worst pain intensity rating of less than 2/10.
Time Frame: Approximately 6 days
Population: Analysis Population consists of 233 participants. 28 out of 261 randomized participants were excluded due to criteria related to the safety of propranolol administration (eg, abnormal ECG findings) or a candidate not being able to complete the study (eg, change in time commitment). These post-randomization exclusions were made for safety reasons and participants were excluded prior to any baseline data collection, induction of exercise-induced muscle injury, and treatment allocation.
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D)
Number analyzed (Participants) | 62 | 57 | 57 | 57
Participants | 39 | 32 | 32 | 32

2. Secondary Outcome: Brief Pain Inventory (BPI) for Pain Duration
Description: The Brief Pain Inventory (BPI) consists of rating pain intensity on an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain intensity imaginable). BPI will be recorded daily and the recovery criterion used for this study will be a BPI rating of current pain 0/10 and worst pain rating of less than 2/10. The pain duration is number of days from the date of induced pain to date of recovery. The longer the duration means a worse outcome.
Time Frame: Daily until recovery criterion met, approximately 5-15 days
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D)
Number analyzed (Participants) | 62 | 57 | 57 | 57
days | 4 [4 to 9] | 4 [1 to 11] | 4 [0 to 11] | 4 [4 to 9]

3. Secondary Outcome: Brief Pain Inventory (BPI) for Worst Shoulder Pain Intensity (Highest Daily Pain Intensity Rating) Recorded During Recovery.
Description: The Brief Pain Inventory (BPI) which consists of rating pain intensity on an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain intensity imaginable). Participants will rate their current, best, and worst pain intensity on the BPI. This measure will be recorded daily through study completion, an average of 5 days. The worst pain intensity rating at Day 2 (when participants usually had the Peak Shoulder Pain Intensity) is reported.
Time Frame: Day 2 value of the worst pain intensity is reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D)
Number analyzed (Participants) | 62 | 57 | 57 | 57
score on a scale | 2.9 (1.9) | 3.2 (2.1) | 2.9 (2.1) | 3.1 (2.0)

4. Secondary Outcome: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH)
Description: The abridged version of the DASH (the QuickDASH) which consists of 11 functional items, with total scores ranging from 0 (not disability) to 100 (complete disability) will be used to assess upper-extremity disability. The primary outcome will be the highest DASH score recorded during the pain intensity recovery period.
Time Frame: Daily until recovery criterion met, approximately 5-15 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D)
Number analyzed (Participants) | 62 | 57 | 57 | 57
score on a scale | 8.2 (8.5) | 10.5 (12.4) | 11.4 (12.9) | 9.4 (8.3)

ADVERSE EVENTS:
Time Frame: 5 days
Description: Mortality and serious adverse events were monitored. Side effects were closely monitored and captured by self-report at the beginning of each study session (starting on day 2), thus reflecting the prior day response to the study drug.
Arm/Group | Personalized Pharmaceutical and Education (C) | Placebo Pharmaceutical, General Education (B) | Placebo Pharmaceutical, Personalized Education (A) | Personalized Pharmaceutical, General Education (D)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/57 | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/57 | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 49/62 | 43/57 | 39/57 | 43/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized Pharmaceutical and Education (C) (N=62) | Placebo Pharmaceutical, General Education (B) (N=57) | Placebo Pharmaceutical, Personalized Education (A) (N=57) | Personalized Pharmaceutical, General Education (D) (N=57)
Light headedness (General disorders) | 17 (22) | 17 (28) | 18 (30) | 14 (17)
Slowed heartbeat (Blood and lymphatic system disorders) | 2 (6) | 4 (4) | 4 (4) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 25 (44) | 24 (56) | 25 (51) | 19 (45)
Fatigue (Musculoskeletal and connective tissue disorders) | 35 (67) | 30 (77) | 32 (87) | 36 (74)
Gastrointestinal upset (Gastrointestinal disorders) | 10 (16) | 11 (18) | 12 (17) | 6 (8)
Allergic reactions (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Dizziness (General disorders) | 6 (6) | 8 (10) | 8 (15) | 8 (11)
Nausea/Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (13) | 7 (12) | 5 (7)
Numbness/tingling in the hands (Nervous system disorders) | 4 (4) | 6 (10) | 6 (9) | 4 (5)
Sleep problems (General disorders) | 12 (21) | 19 (43) | 13 (26) | 14 (33)
Depression (General disorders) | 2 (4) | 2 (4) | 2 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial did not include participants with a clinical conditions. Instead, participants were recruited into this trial and shoulder pain was induced via exercise-induced muscle injury. We then randomly assigned them to 4 different arms, and tested for differences in recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02620579/Prot_SAP_000.pdf